CLINICAL TRIAL: NCT07152587
Title: Randomized, Embedded, Multifactorial, Adaptive Platform Trial of Pathogen-Directed Precision Anti-inflammatory Therapy in Severe Community-Acquired Pneumonia(Core Protocal)
Brief Title: Randomized Adaptive Platform Trial of Pathogen-Directed Anti-inflammatory Therapy in Severe Community-Acquired Pneumonia(Core Protocal)
Acronym: PANDA-SCAP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Qingyuan Zhan (Other)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Director, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-I2M-C&T-B-090
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Severe Community-acquired Pneumonia (sCAP)
Keywords: community-acquired pneumonia; adaptive platform trial; pathogen directed; corticosteroids
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Steroids; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (Placebo Comparator): Receive Standard of care for SCAP, including antibiotics and respiratory support.
  Interventions: Drug: Saline (0.9% NaCl)
- Low dose steroids (Experimental): Intervention: Receive 0.5mg/kg Methylprednisolone
  Interventions: Drug: Low dose steroids
- Moderate dose steroids (Experimental): Intervention: Receive 1.0mg/kg Methylprednisolone
  Interventions: Drug: Moderate dose steroids

INTERVENTIONS:
Drug: Low dose steroids — Receive 0.5mg/kg Methylprednisolone
  Arms: Low dose steroids
Drug: Moderate dose steroids — Receive 1.0mg/kg Methylprednisolone
  Arms: Moderate dose steroids
Drug: Saline (0.9% NaCl) — Saline 100ml
  Arms: Standard of Care

SUMMARY:
Severe community-acquired pneumonia (sCAP) has a high mortality rate of 25-50%. Excessive host inflammatory responses contribute to poor outcomes. Corticosteroid therapy may provide benefit; however, the optimal dosage remains unclear, and it is uncertain whether all etiologies (e.g., Pneumocystis jirovecii, adenovirus, influenza) of sCAP can benefit equally.

This study will first establish a comprehensive trial platform based on a prospective sCAP cohort, embedding a randomized, multifactorial, adaptive platform trial (APT). The response-adaptive design will increase the likelihood of patients being assigned to more effective treatment arms, while Bayesian statistical modeling will dynamically assess the efficacy of interventions, allowing early achievement of study endpoints.

At the starting stage, two pathogen-specific APTs will be conducted, focusing on adenovirus- and pneumocystis Jirovecii-induced sCAP. Patients admitted to the ICU with confirmed diagnoses of adenovirus or pneumocystis Jirovecii-associated sCAP will be randomized into a control group or one of two corticosteroid dosage groups. The primary endpoint will be 28-day all-cause mortality. Completion of these APTs will provide a theoretical basis for novel anti-inflammatory strategies in sCAP.

Moreover, this platform will serve as an essential research infrastructure for the efficient evaluation of new therapeutic options in the event of emerging or re-emerging respiratory pathogens causing sCAP in the future.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU;

  * Age ≥ 18 years;

    * ICU length of stay ≤ 48 hours; ④ Meeting the IDSA/ATS diagnostic criteria for SCAP.

Exclusion Criteria:

* Confirmed diagnosis of hospital-acquired pneumonia (HAP) or ventilator-associated pneumonia (VAP);

  * Expected death within 24 hours;

    * Presence of septic shock prior to randomization; ④ History of allergy or contraindications to corticosteroids (e.g., active gastrointestinal bleeding, severe osteoporosis, uncontrolled hyperglycemia, bone marrow suppression);

      * Active fungal (except Pneumocystis jirovecii), tuberculosis, or hepatitis infection;

        * Receiving ongoing corticosteroid therapy at a dose equivalent to prednisone > 1 mg/kg/day due to underlying disease; ⑦ Participation in this trial within the past 90 days; ⑧ Refusal to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | 28 days from inclusion
  death at 28th day after inclusion

IPD SHARING:
Plan to Share IPD: Undecided